CLINICAL TRIAL: NCT00362674
Title: An Open-label, Observation Study to Evaluate the Durability of Antiviral Activity in Chronic Hepatitis B Patients Who Showed Complete Response in L-FMAU-301,L-FMAU-302 or L-FMAU-303 Trial
Brief Title: Durability of Antiviral Activity in Chronic HBV Patients Who Showed Complete Response in L-FMAU-301,302 or 303 Trial
Status: Completed | Type: Observational
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Hun Jun Jang, Bukwang Pharm.
Other Study IDs: CLV-304
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the durability of antiviral activity in chronic hepatitis B patients who showed complete response in L-FMAU-301,L-FMAU-302 or L-FMAU-303 trial.

ELIGIBILITY:
Inclusion Criteria:

1. The patients who have completed L-FMAU-301, L-FMAU-302 or L-FMAU-303.
2. Patients who have showed complete response (ALT normalization and HBV DNA <4,700 copies/mL in L-FMAU-301 or L-FMAU-302, in addition, HBeAg seroconverted to anti-HBe at the last two visits in L-FMAU-301) after completion of L-FMAU-301 or L-FMAU-302 and treated with the clevudine.
3. Patients who have showed complete response (ALT normalization and HBV DNA <4,700 copies/mL, in addition HBeAg seroconverted to anti-HBe at the last two visits who showed HBeAg positiv at baseline) after completion of L-FMAU-303
4. Patients who were able to give written informed consent prior to study start and to comply with the study requirements.
5. Patients with bilirubin levels less than 2.0 mg/dL, prothrombin time of less than 1.7 (INR), and a serum albumin level of at least 3.5 g/dL at the last visit in L-FMAU-301, L-FMAU-302 or L-FMAU-303.

Exclusion Criteria:

1. Patients who have showed complete response but previously treated with placebo in the L-FMAU-301, L-FMAU-302.
2. Patients who were currently receiving antiviral, immunomodulatory or corticosteroid therapy.
3. Patients previously treated with interferon, lamivudine, lobucavir, famciclovir, adefovir or any other investigational nucleoside for HBV infection.
4. Patients with a history of ascites, variceal hemorrhage or hepatic encephalopathy.
5. Patients co-infected with HCV, HDV or HIV.
6. Patients with a liver mass (hemangioma, nodule), biliary diseases except asymptomatic GB stone during the L-FMAU-301, L-FMAU-302 or L-FMAU-303.
7. Patients who were pregnant or breast-feeding.
8. Patients with a significant gastrointestinal, renal, hepatic (decompensated), biliary diseases except asymptomatic GB stone, bronchopulmonary, neurological, cardiovascular, oncologic or allergic disease. The patients with a benign tumor were excluded if judged by an investigator that the continuation of study would be interfered by benign tumor.
9. Patients who were not suitable to the study if judged by an investigator.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: the patients who completed the previous 301, 302 and 303 studies with clevudine
Sampling Method: Non-Probability Sample
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-suk Lee, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (27):
- South Korea (27):
  - Pusan National University Hospital, Ami-dong, Seo-gu, Busan
  - Kosin Medical Center, Amnam-dong, Seo-gu, Busan
  - Yeungnam University Medical Center, Daemyoung-dong, Nam-gu, Daegu
  - Keimyumg University Dongsan Medical Center, Jung-gu,, Daegu
  - Korea University Guro Hospital, Seoul, Guro-gu
  - St. Mercy's Hospital, Bupyoung-dong, Bupyoung-gu, Incheon
  - Inha University Hospital, Sinhung-dong, Jung-gu, Incheon
  - Wonkwang University Hospital, Iksan, Jeollabuk-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Seoul National University Hospital, Seoul, Jongno-Gu
  - National Cancer Center, Ilsan-gu, Kyounggi-do
  - St. Holly Family Mary's Hospital, Pucheon, Kyounggi-do
  - Pochon CHA University Hospital, Seongnam-gu, Kyounggi-do
  - Gil Medical Center, Incheon, Namdong-Gu
  - Nowon Eulji Hospital, Hagyeil-tong, Nowon-gu, Seoul
  - Korea University Anam Hospital, Anam-dong, Sungbuk-ku, Seoul
  - Kangnam Sacred Heart Hospital, Daelim-dong, Yongdeungpo-gu, Seoul
  - Yongdong Severance Hospital, Dogok-dong, Kangnam-gu, Seoul
  - Korea Cancer Center Hospital, Gongneung-dong, Nowon-gu, Seoul
  - Samsung Medical Center, Ilwon-dong, Songpa-gu, Seoul
  - Seoul Paik Hospital, Jeo-dong, Seoul
  - Ehwa Womans University Mokdong Hospital, Mok-dong, Yangcheon-gu, Seoul
  - Seoul Asan Medical Center, Pungnap-dong, Kangnam-gu, Seoul
  - Kangbuk Samsung Hospital, Pyoung-dong, Chongro-gu,, Seoul
  - Severance Hospital, Shinchon- Dong, Seodaemun-gu, Seoul
  - St. Vincent's Hospital, Ji-dong,, Paldal-gu, Suwon
  - St. Mary's Hospital, Seoul, Yungdungpo-Gu